CLINICAL TRIAL: NCT06065735
Title: An Open-Label, Single Arm, Dose Escalating Concentration-QT Study to Investigate the Cardiac Effects and Safety of Paroxetine in Healthy Adult Participants
Brief Title: Concentration-QT Study of Paroxetine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 219882
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Anxiety Disorders
Keywords: Dose escalation; QTc Interval; Paroxetine; Healthy Adults
MeSH Terms: conditions — Anxiety Disorders | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paroxetine (Experimental)
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine — Paroxetine will be administered

SUMMARY:
The primary purpose of the study is to evaluate the potential effect of paroxetine on QTc interval following escalating doses in healthy participants. Participants with no history of cardiac abnormalities or mood disorders will be enrolled. During the study, participants will take paroxetine at three incremental dose levels. Participants will attend the clinic at screening, baseline, at the end of each dose level administration week, and a final study exit visit. While on treatment outside of clinic visits, participants will be followed-up via video-call. A concentration-QTc analysis will assess any potential correlation between paroxetine plasma concentration and QTc prolongation. In addition, the occurrence of any side-effects will be compared between on and off treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants, both male and female, aged between 18 to 65 years, at the time of signing the informed consent.
* Participants determined as healthy based on medical evaluation by an experienced physician.
* A female participant is eligible to participate if she is of:

  * Nonchildbearing potential defined as premenopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea.
  * Child-bearing potential and agrees to use one of the contraception methods for an appropriate time as mentioned in the study protocol.
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase, and bilirubin ≤ 1.5x (Upper Limit of Normal) ULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Body weight ≥ 45 kilogram (kg) and Body Mass Index (BMI) within the range 18 to 29.5 kilogram per metre square (kg/m2) (inclusive).
* No significant abnormality on 12-lead Electrocardiogram (ECG) at Screening in supine position, including the following specific requirements:

  1. Heart rate ≥ 40 beats per minute
  2. PR interval ≤ 220 milliseconds (msec) (For PR, QRS and QTcF interval, and Q wave, the mean of triplicate ECGs will be used)
  3. Q waves < 50 msec (For PR, QRS and QTcF interval, and Q wave, the mean of triplicate ECGs will be used)
  4. QRS interval to be ≥ 60msec and < 120msec (For PR, QRS and QTcF interval, and Q wave, the mean of triplicate ECGs will be used)
  5. The waveforms must enable the QT interval to be clearly defined
  6. QTcF interval must be < 450msec (machine or manual reading).
* A signed and dated written informed consent obtained from participants capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked) or light smokers (less than 5 cigarettes per day).

Exclusion Criteria:

* History or presence of any medically significant disease that may cause additional risk or interfere with the study procedures or outcome.
* History of symptomatic arrhythmias.
* History of hypersensitivity to paroxetine and excipients
* History of abnormal coagulation parameters, bleeding disorders or conditions which may predispose to bleeding.
* History of, or active suicidal ideation. Includes assessment using the Columbia Suicide Severity Rating Scale (C-SSRS)
* Must not have a pre-diagnosed mood disorder
* Participant is mentally or legally incapacitated.
* A supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHG) at Screening.
* A supine heart rate outside the range 50-90 beats per minute (bpm) at Screening.
* A positive screening Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones).
* A positive drug/alcohol screen at screening or prior to dosing.
* A positive test for Human Immune Virus (HIV) antibody at Screening.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 millilitre [ml]) of beer, 1 glass (125ml) of wine or 1 (25 ml) measure of spirits.
* The participant has participated in a clinical trial and has received an investigational product within the following time prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of the following medications within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of the study medication: monoamine oxidase inhibitors (including linezolid), thioridazine, pimozide, serotonergic drugs (including L-tryptophan, triptans, tramadol, selective serotonin reuptake inhibitors, lithium and fentanyl, tamoxifen, anti-coagulants, clozapine, phenothiazines, tricyclic antidepressants, acetylsalicylic acid, non-steroidal anti-inflammatory drugs, Cox-2 inhibitors, antiarrhythmics, quinolone antibiotics, macrolides (including clarithromycin and erythromycin), ketoconazole and itraconazole
* Use of non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* No current use of any medication other than paracetamol (doses ≤2 grams/day).
* Consumption of Seville oranges, pummelos (members of the grapefruit family) or grapefruit juice from 7 days prior to the first dose of study medication.
* Where participation in the study would result in donation of blood or blood products more than 500 mL within a 3-month period.
* Pregnant females as determined by positive serum β-HCG test at screening or serum/ urine beta-Human chorionic gonadotropin (HCG) prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Participants with unsuitable veins for cannulation and repeat venepuncture.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study investigated the cardiac effects, safety, and tolerability of paroxetine in healthy adult participants.
Pre-assignment Details: A total of 38 participants were enrolled in the study to receive 20 milligrams (mg), 40 mg and 60 mg doses of paroxetine.
Groups:
- Participants Who Received Paroxetine 20 mg: Participants received paroxetine 20 mg tablets, orally once daily from Days 1 to 7.
- Participants Who Received Paroxetine 40 mg: Participants received paroxetine 40 mg tablets, orally once daily from Days 8 to 14.
- Participants Who Received Paroxetine 60 mg: Participants received paroxetine 60 mg tablets, orally once daily from Days 15 to 21.
Period: Paroxetine 20 mg (Days 1 to 7)
Arm/Group | Participants Who Received Paroxetine 20 mg | Participants Who Received Paroxetine 40 mg | Participants Who Received Paroxetine 60 mg
Started | 38 | 0 | 0
Completed | 33 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Paroxetine 40 mg (Days 8 to 14)
Arm/Group | Participants Who Received Paroxetine 20 mg | Participants Who Received Paroxetine 40 mg | Participants Who Received Paroxetine 60 mg
Started | 0 | 33 (Participants who completed 20 mg arm entered 40 mg arm.) | 0
Completed | 0 | 32 | 0
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Paroxetine 60 mg (Days 15 to 21)
Arm/Group | Participants Who Received Paroxetine 20 mg | Participants Who Received Paroxetine 40 mg | Participants Who Received Paroxetine 60 mg
Started | 0 | 0 | 32 (Participants who completed 40 mg arm entered 60 mg arm.)
Completed | 0 | 0 | 31
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants Receiving Paroxetine: Participants received paroxetine tablets titrated to a dose of 60 mg once daily at increments of 20 mg per week. Participants received paroxetine 20 mg tablets, orally once daily from Days 1 to 7 followed by paroxetine 40 mg tablets, orally once daily from Days 8 to 14 and then paroxetine 60 mg tablets orally once daily from Days 15 to 21. Participants were followed-up for up-to Day 48.
Arm/Group | All Study Participants Receiving Paroxetine
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (11.48)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 23
  Female | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race categories (with 0<n<11) are combined into one 'De-identified' category to maintain participant confidentiality and privacy, as they could lead to participant re-identification.
  Participants
    White | 25
    De-identified | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Corrected QT Interval by Fridericia (QTcF Interval)
Description: A standard 12-lead electrocardiogram (ECG) were recorded in a participant using an ECG machine after 10 minutes rest in the supine position. Baseline was defined as the sample obtained on Day -1. Change from Baseline was calculated by subtracting Baseline value from post dose value.
Time Frame: Baseline (Day -1); 0.25 Hours Pre-dose on Day 1; 1, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12 Hours Post-dose on Day 1
Population: Pharmacodynamic Population included all participants in the Safety Population who had at least 1 non-missing ECG assessment. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Participants Who Received Paroxetine 20 mg | Participants Who Received Paroxetine 40 mg | Participants Who Received Paroxetine 60 mg
Number analyzed (Participants) | 33 | 32 | 31
Milliseconds
  0.25 Hours Pre-dose on Day 1 | 1.9 (7.37) | 1.0 (10.82) | 0.9 (9.88)
  1 Hour Post-dose on Day 1 | 2.2 (10.68) | 2.9 (12.60) | 0.6 (13.35)
  2 Hours Post-dose on Day 1 | -3.0 (9.54) | -2.9 (10.83) | -4.2 (11.05)
  3 Hours Post-dose on Day 1 | -7.1 (8.48) | -5.4 (10.10) | -6.9 (8.92)
  4 Hours Post-dose on Day 1 | -4.4 (9.68) | -4.2 (10.48) | -4.6 (10.70)
  4.5 Hours Post-dose on Day 1: number analyzed (Participants) | 33 | 31 | 31
  4.5 Hours Post-dose on Day 1 | -2.5 (8.26) | -1.2 (11.85) | -1.5 (11.15)
  5 Hours Post-dose on Day 1: number analyzed (Participants) | 31 | 32 | 31
  5 Hours Post-dose on Day 1 | -0.3 (10.08) | 0.9 (12.53) | -0.7 (10.37)
  5.5 Hours Post-dose on Day 1 | 4.0 (8.49) | 3.6 (11.91) | 3.2 (10.57)
  6 Hours Post-dose on Day 1 | 4.2 (9.15) | 4.0 (11.35) | 4.7 (8.51)
  8 Hours Post-dose on Day 1 | 1.6 (12.34) | -0.2 (13.35) | -0.1 (11.76)
  10 Hours Post-dose on Day 1 | -5.0 (9.62) | -5.2 (10.22) | -5.0 (12.51)
  12 Hours Post-dose on Day 1 | -0.5 (10.41) | -4.0 (10.61) | -4.2 (12.06)

2. Secondary Outcome: Change From Baseline in Vital Signs: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in the supine position using a semi-automatic blood pressure recording device with an appropriate cuff size after at least 5 minutes of rest. Baseline was defined as the sample obtained on Day -1. Change from Baseline was calculated by subtracting Baseline value from post dose value. Mean and standard deviation (SD) values of vital sign assessments at Day 48 are reported.
Time Frame: Baseline (Day -1) and Day 48
Population: Safety Population included all participants who received at least one dose of study intervention. As all participants received 20, 40 and 60 mg of paroxetine and as there was no intent of comparison of vital signs across these doses, the results were planned to be presented as a single overall arm.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | All Study Participants Receiving Paroxetine
Number analyzed (Participants) | 38
Millimeters of mercury (mmHg)
  Systolic Blood Pressure | 6.474 (5.8713)
  Diastolic Blood Pressure | 4.763 (5.9340)

3. Secondary Outcome: Change From Baseline in Vital Sign: Pulse Rate
Description: Pulse rate was measured in the supine position using a semi-automatic recording device with an appropriate cuff size after at least 5 minutes of rest. Baseline was defined as the sample obtained on Day -1. Change from Baseline was calculated by subtracting Baseline value from post dose value. Mean and SD values of vital sign assessments at Day 48 are reported.
Time Frame: Baseline (Day -1) and Day 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | All Study Participants Receiving Paroxetine
Number analyzed (Participants) | 38
Beats per minute (bpm) | 1.842 (5.0325)

4. Secondary Outcome: Change From Baseline in Vital Sign: Body Temperature
Description: Body temperature measurements were performed in participants. Baseline was defined as the sample obtained on Day -1. Change from Baseline was calculated by subtracting Baseline value from post dose value. Mean and SD values of vital sign assessments at Day 48 are reported.
Time Frame: Baseline (Day -1) and Day 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | All Study Participants Receiving Paroxetine
Number analyzed (Participants) | 38
Degrees Celsius | 0.047 (0.1109)

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose, results in death; was life threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or any other situation as determined per medical and scientific judgment.
Time Frame: Up to Day 48
Population: Safety Population included all participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received Paroxetine 20 mg | Participants Who Received Paroxetine 40 mg | Participants Who Received Paroxetine 60 mg
Number analyzed (Participants) | 38 | 33 | 32
Participants
  AEs | 23 | 19 | 9
  SAEs | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Findings for Hematology, Clinical Chemistry and Coagulation Laboratory Parameters
Description: The laboratory measurements included hematology, clinical chemistry and coagulation parameters. The parameters evaluated were Basophil, Eosinophil, Erythrocyte Mean Corpuscular Volume, Erythrocytes, Hematocrit, Hemoglobin, Lymphocyte, Monocyte, Neutrophils, Platelets, Reticulocytes, Alanine Aminotransferase, Alkaline phosphatase, Aspartate Aminotransferase, Bilirubin, Calcium, Creatinine, Direct Bilirubin, Potassium, Sodium, Creatinine kinase, Prothrombin time (PT), activated partial thromboplastin time (aPTT), international normalized ration (INR). Clinical significance was determined by the investigator. Number of participants with clinically significant findings in hematology, clinical chemistry and coagulation were reported.
Time Frame: Up to Day 48
Population: Safety Population included all participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received Paroxetine 20 mg | Participants Who Received Paroxetine 40 mg | Participants Who Received Paroxetine 60 mg
Number analyzed (Participants) | 38 | 33 | 32
Participants
  Hematology | 0 | 0 | 0
  Clinical chemistry | 0 | 0 | 0
  Coagulation | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Findings for Vital Signs
Description: Vital signs included systolic and diastolic blood pressure, pulse rate and body temperature. Blood pressure and pulse rate were measured with the participant in supine position after at least 5 minutes rest. Clinical significance was determined by the investigator. Number of participants with clinically significant findings in vital signs were reported.
Time Frame: Up to Day 48
Population: Safety Population included all participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received Paroxetine 20 mg | Participants Who Received Paroxetine 40 mg | Participants Who Received Paroxetine 60 mg
Number analyzed (Participants) | 38 | 33 | 32
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Findings for Physical Examinations
Description: Physical examinations included assessment of skin, lungs, cardiovascular system, and abdomen (liver and spleen). Clinical significance was determined by the investigator. Number of Participants with clinically significant findings for physical examinations were reported.
Time Frame: Up to Day 48
Population: Safety Population included all participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received Paroxetine 20 mg | Participants Who Received Paroxetine 40 mg | Participants Who Received Paroxetine 60 mg
Number analyzed (Participants) | 38 | 33 | 32
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and common (>=3%) non-serious adverse events (Non-SAEs) were collected up to Day 48
Description: Safety Population included all participants who received at least one dose of study intervention. AEs were reported Treatment-wise.
Arm/Group | Participants Who Received Paroxetine 20 mg | Participants Who Received Paroxetine 40 mg | Participants Who Received Paroxetine 60 mg
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 23/38 | 19/33 | 9/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Who Received Paroxetine 20 mg (N=38) | Participants Who Received Paroxetine 40 mg (N=33) | Participants Who Received Paroxetine 60 mg (N=32)
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Who Received Paroxetine 20 mg (N=38) | Participants Who Received Paroxetine 40 mg (N=33) | Participants Who Received Paroxetine 60 mg (N=32)
Headache (Nervous system disorders) | 6 | 5 | 2
Somnolence (Nervous system disorders) | 4 | 4 | 1
Dizziness (Nervous system disorders) | 4 | 1 | 0
Disturbance in attention (Nervous system disorders) | 3 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Parosmia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 5 | 3 | 1
Catheter site bruise (General disorders) | 0 | 2 | 0
Catheter site pain (General disorders) | 0 | 1 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 2 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Bruxism (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Dissociation (Psychiatric disorders) | 1 | 0 | 0
Emotional poverty (Psychiatric disorders) | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 2 | 3
Yawning (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 1
Coronavirus infection (Infections and infestations) | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT06065735/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT06065735/SAP_001.pdf